CLINICAL TRIAL: NCT02086513
Title: Phase I Trial of LDE225 for Steroid-refractory Chronic GVHD After Allogeneic HSCT
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Yi-Bin A. Chen, MD, Principal Investigators, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-598
Record Dates: First submitted 2014-03-11; First posted 2014-03-13 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Graft Versus Host Disease
Keywords: Graft versus Host Disease; Allogeneic Stem Cell Transplantation
MeSH Terms: conditions — Graft vs Host Disease | interventions — sonidegib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LDE225 (Experimental): LDE225 will be administered orally, on a continuous once daily dosing schedule at a dose of 200 mg, 400 mg, 600 mg, or 800 mg depending on the specific cohort. Starting dose 200 mg daily for a 28 day cycle. The DLT period will be for the first 2 cycles of therapy. Each cycle is 28 days in length, making the DLT period of minimum of 56 days.
  Interventions: Drug: LDE225

INTERVENTIONS:
Drug: LDE225 — Treatment with LDE225

SUMMARY:
This is a phase I trial of LDE225 for the treatment of steroid-refractory chronic Graft Versus Host Disease (GVHD).

DETAILED DESCRIPTION:
This phase I clinical trial will enroll participants with steroid-refractory chronic GVHD, and likely take approximately 24 months to complete accrual. Treatment will consist of LDE225 given daily for continuous dosing in 28-day cycles. Participants will have undergone allogeneic SCT and have developed chronic GVHD which has not responded sufficiently to systemic corticosteroids (dose of at least 0.25 mg/kg/day of ideal body weight), have relapsed disease while tapering steroids, or not having an adequate response to steroids plus other therapies. Participants who are responding will then be eligible to receive additional courses of therapy. Participants will be followed on trial for 12 months after starting therapy and the trial will be completed when all participants have reached 12 months of follow-up or have withdrawn from the trial.

The initial dose escalation phase of 4 cohorts of participants (each cohort 3-6 participants) will have a primary endpoint of safety and toxicity of administering LDE225 in this setting.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study have to meet all of the following criteria:

* Patients must provide written informed consent prior to any screening procedures.
* Age 18 years or older.
* Recipients of allogeneic hematopoietic cell transplantation (HCT) after either myeloablative or reduced intensity conditioning regimens. Any donor source of stem cells is eligible.
* Participants must be at least 100 days after HCT.
* Patients must have steroid refractory classic cutaneous, myofascial, or sclerodermatous cGVHD (+/- other organ involvement, clinically diagnosed), defined as having persistent signs and symptoms of chronic GVHD despite the use of prednisone at ≥ 0.25 mg/kg/day (or 0.5 mg/kg every other day) for at least 4 weeks in the preceding 12 months (or equivalent dosing of alternate corticosteroids) without complete resolution of signs and symptoms or if not improving on any line of therapy beyond steroids or if treating physician feels that increasing or adding steroids is not in the patient's best interests. Note that the dose of systemic steroids can certainly be lower than 0.25 mg/kg/day at enrollment.
* Stable dose of corticosteroids for 4 weeks prior to enrollment
* No addition or subtraction of other immunosuppressive medications (e.g., calcineurin inhibitors, sirolimus, mycophenolate mofetil) for 4 weeks prior to enrollment. The dose of immunosuppressive medicines may be adjusted based on the therapeutic range of that drug
* ECOG performance status ≤ 3
* Serum Cr ≤ 2 gm / dL
* Adequate hepatic function (total bilirubin < 2.0 mg/dl, AST < 5x ULN), unless hepatic dysfunction is a manifestation of cGVHD. For patients in whom a diagnosis of hemolysis or Gilbert's is made, the total bilirubin is allowed to be elevated. For patients with abnormal LFTs above the thresholds, documented cGVHD on liver biopsy will be required prior to enrollment.
* Patients must have adequate bone marrow function as defined by ANC ≥ 1000 / µl and platelets ≥ 20,000 / µl without growth factor or transfusional support
* Plasma creatine phosphokinase (CK) < 1.5 x ULN
* Patient is able to swallow and retain oral medication

Exclusion Criteria:

* Patients who have had major surgery within 4 weeks of initiation of study medication.
* Patients with concurrent uncontrolled medical conditions that may interfere with their participation in the study or potentially affect the interpretation of the study data.
* Patients unable to take oral drugs or with lack of physical integrity of the upper gastrointestinal tract or known malabsorption syndromes.
* Patients who have previously been treated with systemic LDE225 or with other Hh pathway inhibitors.

  * Patients who have neuromuscular disorders (e.g. inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis and spinal muscular atrophy) or are on concomitant treatment with drugs that are recognized to cause rhabdomyolysis, such as HMG CoA inhibitors (statins), clofibrate and gemfibrozil, and that cannot be discontinued at least 2 weeks prior to starting LDE225 treatment. If it is essential that the patient stays on a statin to control hyperlipidemia, only pravastatin may be used with extra caution.
  * Patients who are planning on embarking on a new strenuous exercise regimen after initiation of study treatment. NB: Muscular activities, such as strenuous exercise, that can result in significant increases in plasma CK levels should be avoided whilst on LDE225 treatment.
* Patients who have taken part in an experimental drug study within 4 weeks or 5 half-lives, whichever is longer, of initiating treatment with LDE225.
* Patients who are receiving other anti-neoplastic therapy (e.g. chemotherapy, targeted therapy or radiotherapy) concurrently or within 2 weeks of starting treatment with LDE225.
* Patients who are receiving treatment with medications known to be strong inhibitors or inducers of CYP3A4/5 or drugs metabolized by CYP2B6 or CYP2C9 that have a narrow therapeutic index, and that cannot be discontinued before starting treatment with LDE225. Medications that are strong CYP3A4/5 inhibitors should be discontinued at least 7 days and strong CYP3A/5 inducers for at least 2 weeks prior to starting treatment with LDE225. Note that patients who require antifungal prophylaxis are preferred to be on fluconazole, and, patients taking voriconazole or posaconazole who must continue are excluded from the dose escalation phase of the study. Once the MTD is established, patients taking voriconazole or posaconazole will be allowed to enroll but at a dose adjustment to be determined before the expansion phase opens.
* Ongoing prednisone requirement > 1 mg/kg/day (or equivalent)
* Exposure to any new immunosuppressive medication in the 4 weeks prior to enrollment.
* ECP therapy within 4 weeks prior to enrollment
* Active disease relapse
* Active, uncontrolled infection
* Impaired cardiac function or clinically significant heart disease, including any one of the following:

  * Angina pectoris within 3 months
  * Acute myocardial infarction within 3 months
  * QTc > 450 msec for males and > 470 msec for females on the screening ECG
  * A past medical history of clinically significant ECG abnormalities or a family history of prolonged QT-interval syndrome
  * Other clinically significant heart disease (e.g. congestive heart failure, uncontrolled hypertension, history of labile hypertension, or history of poor adherence with an antihypertensive regimen)
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/mL).
* Patients who are not willing to apply highly effective contraception during the study and through the duration as defined below after the final dose of study treatment.

  * Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, must use highly effective contraception during the study and through 6 months after the final dose of study treatment. Highly effective contraception is defined as either:
  * Total abstinence: When this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
  * Sterilization: Patient has had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
  * Male partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). [For female study patients, the vasectomized male partner should be the sole partner for that patient]
  * Use a combination of the following (both a+b):

    * Placement of a non-hormonal intrauterine device (IUD) or non-hormonal intrauterine system (IUS)
    * Barrier method of contraception: Condom or Occlusive cap (diaphragm or cervical vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.
    * Note: Hormonal contraception methods (e.g. oral, injected, implanted) are not allowed to count as contraception as it cannot be ruled out that the study drug decreases the effectiveness of hormonal contraception. Patients are able to continue taking oral contraceptives if desired.
    * Note: Woman are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL and estradiol < 20 pg/mL or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential
  * Male patient must use highly effective (double barrier) methods of contraception (e.g., spermicidal gel plus condom) for the entire duration of the study, and continue using contraception and refrain from fathering a child for 6 months following the study drug. A condom is required to be used also by vasectomized men as well as during intercourse with a male partner in order to prevent delivery of the study treatment via seminal fluid
  * Sexually active males who are unwilling to use a condom during intercourse while taking the study drug and for 6 months after stopping investigational medications and agree not to father a child in this period.
* Patients unwilling or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of LDE225 when given as treatment for steroid-refractory chronic GVHD. | 2 years
  Maximum tolerated dose of LDE225 when given as treatment for steroid-refractory chronic GVHD.

SECONDARY OUTCOMES:
Overall Response Rate of LDE225 | 2 Years
  Testing the efficacy of LDE225 for the treatment of steroid-refractory chronic GVHD as described by overall response rate
Incidence of serious infections after starting treatment with LDE225 | 2 Years
  Incidence of serious infections after starting treatment with LDE225
Ability to decrease baseline steroid dose after starting therapy with LDE225 as measured by systemic steroid dosing at 3, 6, and 12 months after starting therapy with LDE225 | 2 Years
  Ability to decrease baseline steroid dose after starting therapy with LDE225 as measured by systemic steroid dosing at 3, 6, and 12 months after starting therapy with LDE225
Assessing patient-reported quality of life at 3 months, 6 months, and 12 months in patients on LDE225 therapy compared to baseline measures prior to study enrollment. | 2 Years
  Assessing patient-reported quality of life at 3 months, 6 months, and 12 months in patients on LDE225 therapy compared to baseline measures prior to study enrollment.
Assessing patient-reported chronic GVHD symptom severity at 3 months, 6 months, and 12 months in patients on LDE225 therapy compared to baseline measures prior to study enrollment. | 2 Years
  Assessing patient-reported chronic GVHD symptom severity at 3 months, 6 months, and 12 months in patients on LDE225 therapy compared to baseline measures prior to study enrollment.
6-month and 12-month cGVHD progression-free survival | 1 Years
  6-month and 12-month cGVHD progression-free survival
6-month and 12-month overall survival | 1 Year
  6-month and 12-month overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Bin Chen, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] DeFilipp Z, Nazarian RM, El-Jawahri A, Li S, Brown J, Del Rio C, Smith M, Valles B, Ballen KK, McAfee SL, Rosenblatt J, Antin JH, Cutler CS, Chen YB. Phase 1 study of the Hedgehog pathway inhibitor sonidegib for steroid-refractory chronic graft-versus-host disease. Blood Adv. 2017 Oct 5;1(22):1919-1922. doi: 10.1182/bloodadvances.2017011239. eCollection 2017 Oct 10. PMID 29296838